CLINICAL TRIAL: NCT01098201
Title: The Effect of Certolizumab on Lower Extremity Lymph Flow in Rheumatoid Arthritis
Brief Title: Certolizumab and Lower Extremity Lymph Flow in Rheumatoid Arthritis (RA)
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Christopher Ritchlin, M.D., M.P.H.; Professor of Medicine Allergy, Immunology & Rheumatology Division, University of Rochester
Other Study IDs: RSRB - 27553
Record Dates: First submitted 2010-03-30; First posted 2010-04-02 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Certolizumab; TNF; RA; Cizmia
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Certolizumab — Subcutaneous administration on a monthly basis for six months
  Other Names: Cizmia

SUMMARY:
This open-label pilot study will select subjects who are inadequate responders to methotrexate. These subjects will receive certolizumab subcutaneously on a monthly basis for six months. The study is attempting to determine the following:

1. Is lymphatic flow altered in the extremities of RA patients with an inflamed knee?
2. Is resolution of synovitis associated with a restoration of lymphatic flow and lymph node volume following therapy with certolizumab?
3. Can Doppler ultrasound be used to detect and follow alterations of lymph node size?

DETAILED DESCRIPTION:
Ten RA subjects with unilateral knee synovitis, who have not responded to methotrexate, will be recruited from our early RA Clinics. Following enrollment, the subjects will have a technetium sulfur colloid scan performed on both lower extremities followed by a baseline 3 Tesla contrast-enhanced magnetic resonance imaging (3T CE-MRI) study and Doppler US on the involved knee as described below. The overall disease activity will be determined by the DAS 28 and activity in the involved knee with the RAOS instrument; an outcome measure that quantifies the degree of tenderness, swelling and function in monoarthritis. The subjects will then receive 18 weeks of certolizumab and three of the ten subjects will undergo repeat technetium sulfur colloid scans. To test our hypotheses, we will select three responders based on the RAOS response. We will select only three of the 10 for repeat nuclear studies because this number of subjects will allow us to test our hypothesis without the need to perform the scan on all the subjects. All ten subjects with have 3T CE-MRI, Doppler US and clinical evaluations performed at the 18 week time point. The subjects will continue on certolizumab for a total of 24 weeks.

Sulfur Colloid Technetium Scan. A nuclear radiology technician will inject 0.25cc of technetium sulfur colloid into the first through third web spaces of the feet in both lower extremities. In healthy controls the transit time from the feet to the aortic bifurcation is about 30 minutes. The transit time of the tracer will be measured in both lower extremities at the knee, inguinal ligament and at the aortic bifurcation. Images will be obtained with a nuclear camera according to standard protocol serially over the first hour and delayed images acquired in 4 to 6 hours if necessary. Three subjects who have responded to certolizumab will have the scan repeated at 18 weeks as outlined above.

3T CE-MRI. Two radiologists will independently quantify LN volume and CE of all nodes in the popliteal area from the MRI. These radiologists will also quantify the extent of synovial inflammation, cartilage erosion and bone marrow edema via the RA MRI scoring system (RAMRIS). Consensus findings will be reached and the volume and CE for each node identified together with the RAMRIS will be entered into a database for this study. At the end of the study, we will assess the trend of anti-TNF therapy on:

1. The number of detectable LN in the popliteal fossa
2. Mean LN volume for detectable LN
3. Mean LNCE for detectable LN
4. LNcap for detectable LN
5. RAMRIS, by plotting the change over 8 weeks for each knee independently as we have previously described for anti-TNF effects on bone marrow edema in PsA subjects. The relationship between LN and clinical response to therapy will be assessed from deriving the significance of the correlation coefficient (x2) of LNcap vs DAS28 respectively, as we have done for bone marrow edema vs. DAS28 in PsA subjects on anti-TNF therapy.

Doppler US. Ultrasound examinations of PLN will be obtained at baseline and 18 weeks after anti-TNF therapy as follows. All US examinations will be performed by a rheumatologist (RT) certified in musculoskeletal ultrasound.

All subjects will be examined sonographically for the presence of inflammatory changes in the knee joint. The involved knee will be examined sonographically for the presence of the following:

1. Effusion. A distension of pre-femoral and suprapatellar fat pads of >4.8 mm will be noted as an effusion in the suprapatellar recess of the knee joint.
2. Synovial thickening. Hypoechoic, often nodular or villous appearing tissue within the suprapatellar recess that is distinct from the hyperechoic capsular structures and prefemoral and suprapatellar fat pads will be noted as synovitis.
3. Synovial hyperemia. If proliferative synovial tissue is identified, this tissue will be examined with Doppler ultrasound for the presence of increased blood flow. This will be defined as the presence of color pixels in such synovial tissue that appear in synchronicity with the subject's pulse.

In all subjects, affected joints will be examined with gray scale and Doppler ultrasound. Affected joints will be examined sonographically for the presence of the following:

1. Effusion in a joint will be defined as a hypoechoic area within the hyperechoic joint capsule. Such anechoic intra-articular fluid will be displaceable by pressure of the US probe. This helps distinguish joint fluid from intra-articular hyaline cartilage, which is also anechoic to hypoechoic in appearance but is not displaceable by pressure of the probe. The distension of the joint capsule will be measured using sonographic calipers. This distension will be compared with normal values to assess the degree of effusion.
2. Synovial thickening. The synovial lining cells are only one to three cell layers strong in an unaffected joint, so intra-articular, hypoechoic proliferative synovial tissue can be readily distinguished sonographically from more hyperechoic capsular structures. Thickening, if present, will be measured using sonographic calipers.
3. Synovial hyperemia. If synovial thickening is detected, this tissue will be examined sonographically for the presence of Doppler flow as a measure of hyperemia and inflammation.
4. Bony erosions. Erosions will be defined as breaks in the cortical bony contour seen in two perpendicular planes.

The dimensions of all the PLN that can be imaged and cataloged for longitudinal analysis. Synovitis and erosions will also be scored by ultrasound before and after therapy.

Outcome Measures:

1. Technetium sulfur colloid scan

   1. The primary outcome measure for this study is the transit time from foot to the umbilicus (T3) after injection of radioisotope in the limb with the inflamed knee compared to the transit times (T3) in the extremity of the uninflamed knee.
   2. Secondary outcome measures are:

      * the transit times from the foot to the knee (T1) and inguinal ligament (T2) of the radioisotope in both lower extremities
      * Intensity of counts (intensity/area of interest) in the knee, inguinal ligament and umbilicus in both lower extremities.
      * Change in transit times and tracer intensity in the three sites after 12 weeks of certolizumab treatment in the involved extremity (3 subjects only)
2. MRI (secondary):

   1. The amount of contrast enhancement and volume of the draining PLN will be analyzed before and 18 weeks after treatment with certolizumab.
   2. The amount of synovitis, joint effusion, erosion and bone marrow edema will be quantified using the RAMRIS scoring system before and 18 weeks after treatment.
3. Doppler ultrasound (secondary):

   1. Number of detectable LN in the popliteal fossa.
   2. Mean LN size (maximum area).
   3. Secondary measures: synovitis, joint effusion, erosions, and blood flow will also be assessed in the involved joint.
4. Clinical Assessments:

   1. Degree of tenderness (0-3) with subject visual analogue scale (VAS) and swelling with MD VAS (0-3) of the inflamed before and after treatment.
   2. Rheumatoid Arthritis Outcome Score (RAOS)before and after treatment.
   3. Disease Activity Score (DAS 28) score to assess overall joint response to therapy with certolizumab

ELIGIBILITY:
Inclusion

* Inflammatory arthritis. Patients with RA according to the American College of Rheumatology criteria.
* Inadequate response to treatment following 3 months of methotrexate (15-20 mg per week). Inadequate response will be defined as the presence of knee inflammation and at least 2 active joints. If the knee has an effusion, fluid must be obtained to exclude infection or crystalline disease.
* Knee inflammation in one knee determined on physical exam and confirmed by Doppler ultrasound. We will include patients with bilateral knee inflammation only if one knee is more inflamed than the contralateral knee. The comparative level of inflammation will be determined by clinical examination and Doppler US.
* Patients must be willing to undergo a sulfur colloid technetium scan, knee ultrasound and MRI of the knee.

Exclusion Criteria

* Contra-indication to anti-TNF agent.
* History of recurrent infections.
* Prosthetic knee joint
* Recent surgery or trauma to a knee joint
* Lymphedema
* Lymphoproliferative disorder
* Claustrophobia such that they cannot undergo an MRI of the knee
* GFR<60 cc/min
* Morbid obesity
* Foot disease: active ankle or forefoot synovitis, recent trauma, cellulitis or edema.
* Peripheral vascular disease
* Diabetes
* Active skin inflammation in the lower extremities
* Solid Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female RA sufferers not less than 18 yrs of age who are currently experiencing knee synovitis. Racial and ethnic origin of subjects will be monitored to reflect the diversity of our community.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2010-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Initial lymphatic flow in inflamed knee | Week 0 (initial medication dose)
  To examine the lymph flow in the knee joint of RA patients before therapy with certolizumab using technetium sulfur colloid scans, MRI and Doppler ultrasound.
Initial synovitis and its association with lymph flow and node volume | Week 0 (initial medication dose)
  To examine lymph flow and lymph node volume before therapy with certolizumab. Flow volume will be assessed using technetium sulfur colloid scans while lymph node volume will be assessed using MRI.
Initial Doppler ultrasound assessment of lymph node size | Week 0 (initial medication dose)
  To assess lymph node volume before therapy with certolizumab.
Post medication lymphatic flow in inflamed knee | Wk 18
  To examine lymph flow in the knee joint of RA patients after therapy with certolizumab using technetium sulfur colloid scans, MRI and Doppler ultrasound
Post medication synovitis and its association with lymph flow and node volume | Wk 18
  To examine lymph flow and lymph node volume after therapy with certolizumab. Flow volume will be assesses using tecnetium sulfur colloid scan while lymph node volume will be assessed using MRI.
Post medication Doppler ultrasound assessment of lymph node size | Wk 18
  To assess lymph node volume after therapy with certolizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ritchlin, MD / MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Rahimi H, Bell R, Bouta EM, Wood RW, Xing L, Ritchlin CT, Schwarz EM. Lymphatic imaging to assess rheumatoid flare: mechanistic insights and biomarker potential. Arthritis Res Ther. 2016 Sep 1;18:194. doi: 10.1186/s13075-016-1092-0. PMID 27586634
- [Derived] Li J, Zhou Q, Wood RW, Kuzin I, Bottaro A, Ritchlin CT, Xing L, Schwarz EM. CD23(+)/CD21(hi) B-cell translocation and ipsilateral lymph node collapse is associated with asymmetric arthritic flare in TNF-Tg mice. Arthritis Res Ther. 2011 Aug 31;13(4):R138. doi: 10.1186/ar3452. PMID 21884592